CLINICAL TRIAL: NCT06917287
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Design Clinical Study to Evaluate the Efficacy of Native CT-II® in Individuals With Knee Osteoarthritis
Brief Title: A Clinical Study to Evaluate the Efficacy of Native CT-II® in Individuals With Knee Osteoarthritis
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Vedic Lifesciences Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 241001/NCTII/OA
Record Dates: First submitted 2025-04-01; First posted 2025-04-08 (Actual); Last update posted 2026-01-22 (Actual); Status verified 2026-01

CONDITIONS: Knee Osteoarthritis (OA)
MeSH Terms: conditions — Osteoarthritis, Knee | interventions — Glucosamine; Chondroitin; microcrystalline cellulose

STUDY DESIGN:
Intervention Model Description: Randomized, double-blind, placebo-controlled, parallel design
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Native CT-II® (undenatured type II collagen) (Experimental): Strength: 40 mg in 3 capsules
  Dose Regimen:
  3 yellow capsules containing MCC after breakfast with water 3 blue capsules containing 40 mg Native CT-II® & MCC after dinner with water Route of administration: Oral
  Interventions: Dietary Supplement: Native CT-II® (undenatured type II collagen)
- Glucosamine HCL + Chondroitin Sulphate (G+C) [Comparator] (Active Comparator): Strength: 2700 mg (1500 mg G + 1200 mg C)
  Dose Regimen:
  3 yellow capsules containing G+C after breakfast with water 3 blue capsules containing G+C after dinner with water Route of administration: Oral
  Interventions: Dietary Supplement: Glucosamine HCL + Chondroitin Sulphate (G+C) [Comparator]
- Placebo [Microcrystalline Cellulose (MCC)] (Placebo Comparator): Strength: 2700 mg excipient
  Dose Regimen:
  3 yellow capsules containing MCC after breakfast with water 3 blue capsules containing MCC after dinner with water Route of administration: Oral
  Interventions: Dietary Supplement: Placebo [Microcrystalline Cellulose (MCC)

INTERVENTIONS:
Dietary Supplement: Native CT-II® (undenatured type II collagen) — Strength: 40 mg in 3 capsules
  Dose Regimen:
  3 yellow capsules containing MCC after breakfast with water 3 blue capsules containing 40 mg Native CT-II® & MCC after dinner with water Route of administration: Oral
  Arms: Native CT-II® (undenatured type II collagen)
Dietary Supplement: Glucosamine HCL + Chondroitin Sulphate (G+C) [Comparator] — 2700 mg (1500 mg G + 1200 mg C) 3 yellow capsules containing G+C orally after breakfast with water & 3 blue capsules containing G+C after dinner with water
  Arms: Glucosamine HCL + Chondroitin Sulphate (G+C) [Comparator]
Dietary Supplement: Placebo [Microcrystalline Cellulose (MCC) — 2700 mg excipient 3 yellow capsules containing MCC orally after breakfast with water 3 blue capsules containing MCC after dinner with water.
  Arms: Placebo [Microcrystalline Cellulose (MCC)]

SUMMARY:
This randomized, double-blind, placebo-controlled clinical study evaluates the efficacy of Native CT-II® (undenatured type II collagen) in individuals with knee osteoarthritis using a parallel design.Participants are assigned to one of three groups:

Group 1 receives Native CT-II® (40 mg daily individed doses), Group 2 receives Glucosamine HCL + Chondroitin Sulphate (2700 mg daily as acomparator), and Group 3 receives a placebo (Microcrystalline Cellulose). All participants take threecapsules after breakfast and three after dinner for 90 days . The study aims to screen approximately 142 participants

, randomizing around 114 (considering a 20% dropout rate), with a target of 90completed participants (30 per group). Osteoarthritis (OA) is a degenerative joint disorder causing pain, stiffness, and reduced mobility,primarily affecting older adults. It is a leading cause of disability, with knee OA being the mostprevalent form. The global burden of OA is rising due to aging populations and increasing obesityrates, necessitating improved treatment options. Current management focuses on symptom reliefthrough non-pharmacological (exercise, weight loss) and pharmacological (NSAIDs, analgesics)interventions, though these can have adverse effects.

Undenatured type II collagen (NCTII), derived from chicken sternum, has emerged as a potentialsupplement for joint health. It triggers an immune response that reduces inflammation and supportscartilage repair. Clinical studies show that NCTII improves joint function, pain, and quality of life,outperforming glucosamine and chondroitin with fewer side effects. A new study aims to evaluatethe efficacy of Native CT-II® in individuals with Grade II and III knee OA over 90 days, comparing itto glucosamine-chondroitin and placebo groups.

ELIGIBILITY:
Inclusion Criteria:

* 1.Individuals ready to give voluntary, written informed consent to participate in the study.

  2.Males and females of age between 40 to 65 years (including both values) suffering from Knee Osteoarthritis under no medications.

  3.Body mass index (BMI) between 18.5 to 29.9 kg/m2 (including both values). 4.mWOMAC total score ≥ 75. 5. Individuals with knee pain having VAS score of greater than or equal to 60 mm on a 100 mm VAS scale.

  6.Radiographic evidence (lateral and anterio-posterior weight-bearing standing X-ray) of grade II/III (in 2: 1 ratio) knee Osteoarthritis (OA) for index joint (The knee with the higher pain score will be designated as the index joint for the study) based on the Kellgren and Lawrence (K&L) radiographic entry criteria for OA -
  * Grade II: Possible joint space narrowing (JSN) with definite osteophyte formation.
  * Grade III: Definite joint space narrowing, multiple osteophyte formations, some sclerosis, and possible deformity of bony ends.

    7.Individuals with a history of symptomatic knee joint pain of at least 3 months.

    8.Non-vegetarians (regardless of whether they eat chicken, fish, goat mutton, pork, beef or eggs) 9.Willing to abstain from food (fish, meat, bone broth, eggs, etc) containing Type II collagen from cartilage 48 h before all assessment visits.

    10.Willing to stop using rescue medication 48 hours prior to every assessment visits.

    11.Willing to stop the restricted dietary supplements, home-based remedies, and any other form of topical products or medications (mainly includes NSAIDs and local analgesics, DMARD, corticosteroids, etc) for knee joint pain relief or any other reason for the entire study duration.

(Note: only hot and cold fomentation will be allowed, and the participant has to record the daily frequency of fomentation in the diary. The hot/cold fomentation needs to be stopped 48 hours prior to all assessment visits.).

12.Individuals using the western toilet at home and/or workplace. 13.Willing to abstain from alcohol, caffeine, and vigorous physical activity for 24 hours before every study visit.

14.Willingness to participate and comply with the study procedures and required visits.

Exclusion Criteria:

* 1.Individuals who have been injured near the knee joint region in the past six months.

  2.Individuals with a history of knee surgery, replacement or any non-knee surgical procedures that may impact the study outcomes.

  3.Individuals who have used intra-articular injections, platelet replacement therapy, stem cell therapy and or steroids for joint health issues in the last six months.

  4.Individuals who have any other chronic disease or condition, or inflammatory disease conditions and/ or are using any medication or dietary supplements or ayurvedic medications or topical ointment/oil/gel for joint health that in the judgment of the Investigator would put the individual at unacceptable risk for an individual in the study or may interfere with evaluations in the study or noncompliance with treatment or visits.

  5.History or presence of clinically significant renal, hepatic, endocrine, biliary, gastrointestinal, pancreatic, or neurological disorders, that in the judgment of the Investigator, would interfere with the individual's ability to provide informed consent, comply with the study protocol (which might confound the interpretation of the study results), or put the individual at undue risk.

  6.History of uncontrolled hypertension and/or systolic blood pressure more than or equal to 140 mmHg and/or diastolic blood pressure more than or equal to 90 mmHg.

  7.Fasting blood glucose (FBG) more than or equal to 126 mg/dl 8.Known cases of gout and/or hyperuricemia 9.Any history or evidence of allergy to chicken, shellfish, eggs or protein products in the past.

  10.Use of collagen supplements (as dietary supplements) 11.History of bleeding disorders (e.g. Hemophilia, sickle cell anemia) 12.Other pathologic lesions on X-ray of the knee. 13.Any other condition that would prohibit completion of the exercise protocols.

  14.Individuals who have participated in a clinical study with an Investigational product within 90 days before pre-screening, and who plan to participate in another study during the study period.

  15.Not willing to abstain from the use of NSAIDs (including aspirin 50 mg/day for cardiovascular health).

  16.Pregnant or Lactating females. 17.Individuals having a history of drug or alcohol abuse. 18.Current smokers

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 114 (Estimated)
Dates: Start 2025-04-20 (Actual); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-02-15 (Estimated)

PRIMARY OUTCOMES:
To evaluate the effect of consumption of Native CT-II on knee joint health asassessed by change in modified Western Ontario and McMaster UniversityOsteoarthritis Index total score as compared to baseline,Glucosamine HCL + Chondroitin Sulphate an | day 0, day 7, day 30, day 60 and day 90
  The primary efficacy variable for this study is the total mWOMAC index score. The scores from each subscale will be combined, with the pain subscale ranging from 0 to 20, the stiffness subscale from 0 to 8, and the physical function subscale from 0 to 80. Participants with knee OA will complete the mWOMAC index total score.

SECONDARY OUTCOMES:
To assess the effect of Native CT-II® in comparison to baseline, GlucosamineHCL + Chondroitin Sulphate and placebo on Knee joint pain as assessed bychange in mWOMAC - Pain subscale (mWOMAC-P) score. | day 0, day 7, day 30, day 60 and day 90
  The pain subscale (mWOMAC-P) of the mWOMAC index consists of 5 questions that assess the level of pain experienced by individuals with OA in the index joint. Responses are recorded using a 5-point likert scale, where higher scores correspond to greater pain. The scale ranges from 0 ("No pain") to 4 ("Extreme pain"), with the total score for mWOMAC-P ranging from 0 to 20. Participants with knee OA will complete the mWOMAC-P.
To assess the effect of Native CT-II in comparison to baseline, GlucosamineHCL + Chondroitin Sulphate and placebo on Knee joint stiffness as assessedby change in mWOMAC - Stiffness subscale (mWOMAC-S) score. | day 0, day 7, day 30, day 60 and day 90
  The stiffness subscale (mWOMAC-S) of the mWOMAC index consists of 2 questions that assess the level of stiffness in the index joint, characterized by resistance to movement, along with pain and discomfort. Responses are recorded using a 5-point likert scale, where higher scores indicate greater stiffness. The scale ranges from 0 ("No stiffness") to 4 ("Extreme stiffness"), with the total score for mWOMAC-S ranging from 0 to 8. Participants with knee OA will complete the mWOMAC-S on day 0, day 7, day 30, day 60 and day 90 using the e-diary.
To assess the effect of Native CT-II in comparison to baseline, GlucosamineHCL + Chondroitin Sulphate and placebo on Knee joint function as assessedby change in mWOMAC - Physical Function subscale (mWOMAC-PF) score. | Day 0, Day 7, Day 30, Day 60, and Day 90
  The physical function subscale (mWOMAC-PF) of the mWOMAC index consists of 20 questions assessing the level of difficulty experienced in the index joint due to OA. Responses are recorded on a 5-point likert scale, where higher scores reflect greater functional impairment. The scale ranges from 0 ("No difficulty") to 4 ("Extreme difficulty"), with the total possible score for mWOMAC-PF ranging from 0 to 80. Participants with knee OA will complete the mWOMAC-PF.
To assess the effect of Native CT-II in comparison to baseline, GlucosamineHCL + Chondroitin Sulphate and placebo on acute knee joint pain assessedby change on 100 mm Visual Analogue Scale. | Day 0, Day 7, Day30, Day 60 and 90
  The pain VAS is a tool used to assess pain intensity. It consists of a 100 mm line with two endpoints representing the extremes of pain, such as "no pain" at one end and "extreme pain" at the other.40 It is reliable and valid measure for measuring acute pain.41 Participants will rate their pain by marking a point along the line that reflects their pain level.
To assess the effect of Native CT-II in comparison to baseline, GlucosamineHCL + Chondroitin Sulphate and placebo on Knee pain and functions asassessed by change in knee Injury and Osteoarthritis Outcome Score. | Day 0, Day 7, Day30, Day 60 and 90
  The Knee Injury and Osteoarthritis Outcome Score (KOOS) questionnaire is a self-administered tool designed to evaluate both short- and long-term outcomes relevant to individuals following a knee injury and pain. It measures five key domains: pain, symptoms, activities of daily living, sports and recreational function, and knee-related quality of life. The KOOS meets standard criteria for outcome measures, making it suitable for tracking the progression of knee injuries and the effectiveness of treatments.
To assess the effect of Native CT-II in comparison to baseline, GlucosamineHCL + Chondroitin Sulphate and placebo on Average number of rescuemedication taken by participants in each group. | Day 0, Day 7, Day30, Day 60 and 90
  Rescue medication use will be evaluated by counting the number of tablets consumed against the number of tablets dispensed at each of the visits for each study. An average number of rescue medications taken by participants in each group will be recorded and will be compared across the groups
To assess the effect of Native CT-II in comparison to baseline, GlucosamineHCL + Chondroitin Sulphate and placebo on Severity of osteoarthritis asassessed by change in Lequesne Functional Index test score. | Day 0, Day 7, Day30, Day 60 and 90
  Participants will self-administer the questionnaire via an e-diary on days 0, 7, 30, 60, and 90. They must avoid rescue medication and hot/cold fomentation for 48 hours before clinic visits. The knee with the highest pain score is designated as the index joint. Questions have graded options reflecting severity, with subscale scores ranging from 0 to 8, leading to a total LFI score between 0 and 24.48. A higher score indicates greater joint severity.

CONTACTS AND LOCATIONS:
Locations (5):
- India (5):
  - Proactive Othopedic Clinic, Mumbai, Maharashtra
  - Ayush Nursing Home, Mumbai, Maharashtra
  - Diamond Orthopedic & Multispeciality Hospital, Mumbai, Maharashtra
  - O2 Clinic, Nashik, Maharashtra
  - Sparsh Superspeciality Hospital, Panvel, Maharashtra

IPD SHARING:
Plan to Share IPD: No